CLINICAL TRIAL: NCT01605721
Title: Efficacy and Safety of Xience in Coronary arEry Disease aLL-comers After stENTing Using the PRIME Platform (EXCELLENT-PRIME Registry)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Hyo-Soo Kim, MD PhD, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1101-054-347
Record Dates: First submitted 2011-07-18; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Artery Disease
Keywords: Everolimus; XIENCE PRIME; Drug eluting stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- XIENCE PRIMETM everolimus-eluting coronary stent (Experimental)
  Interventions: Device: XIENCE PRIMETM everolimus-eluting coronary stent

INTERVENTIONS:
Device: XIENCE PRIMETM everolimus-eluting coronary stent — Active prospective registration of patients receiving the following stent
  : XIENCE PRIMETM

SUMMARY:
Objectives:

1. To evaluate the safety and long-term effectiveness of coronary stenting with the XIENCE PRIMETM in a cohort of "real world" patients and lesion subsets.
2. To determine clinical device and procedural success during commercial use of XIENCE PRIMETM coronary stent

Study population : Approximately consecutive 2000 patients treated with XIENCE PRIMETM

Study period

* Patient enrollment: 2011.05 ~ 2012.04
* End of follow-up period: 2015. 02 (3 years of follow-up)

Primary endpoint

: Target Lesion Failure (TLF) rate at 12 months

Secondary endpoint:

* In-stent & In-segment Late Loss at 9 months
* Stent Thrombosis at 24 hours (acute), 30 days (subacute), 1 year (late), yearly up to 3 years (very late)
* Target Vessel Failure at 12 months (composite of cardiac death, MI, and TVR)
* Any death, cardiac death, MI, TLR, TVR at 30 days, 9months, 1 year, 3 years
* Composite rate of cardiac death and any MI up to 3 years
* Composite rate of all death and any MI up to 3 years
* Composite rate of all death, any MI (Q-wave and non Q-wave) and any repeat revascularization up to 3 years
* Compliance and therapy interruptions with prescribed adjunctive antiplatelet therapy up to 3 years
* Procedural success up to 1 day
* Angiographic success up to 1 day

ELIGIBILITY:
Inclusion Criteria

* The patient agrees to participate in this study by signing the informed consent form. Alternatively, a legally authorized patient representative may agree to the patient's participation in this study and sign the informed consent form.

Angiographic Inclusion Criteria

* There are no angiographic inclusion criteria for this study.

Exclusion criteria

* There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) rate at 12 months | 12 months

SECONDARY OUTCOMES:
In-stent & In-segment Late Loss at 9 months | 9 months
Stent Thrombosis at 24 hours (acute), 30 days (subacute), 1 year (late), yearly up to 3 years (very late) | 24 hours, 30 days, up to 3 years
Any death, cardiac death, MI, TLR, TVR at 30 days, 9 months, 1 year, 3 years | 30 days, 9 months, 1 year, up to 3 years
Composite rate of cardiac death and any MI up to 3 years | up to 3 years
Composite rate of all death and any MI up to 3 years | up to 3 years
Composite rate of all death, any MI (Q-wave and non Q-wave) and any repeat revascularization up to 3 years | up to 3 years
Compliance and therapy interruptions with prescribed adjunctive antiplatelet therapy up to 3 years | up to 3 years
procedural success up to 1 day | 1 day
  failure : CK-MB of >3 times the upper limit of normal
angiographic success up to 1 day | 1 day
  success : a minimum stenosis diameter reduction to <20% in the presence of grade 3 TIMI flow (assessed by angiography)

CONTACTS AND LOCATIONS:
Overall Officials: Hyo-Soo Kim, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kang J, Han JK, Kang DY, Zheng C, Yang HM, Park KW, Kang HJ, Koo BK, Kim HS. SYNTAX Score and SYNTAX Score II Can Predict the Clinical Outcomes of Patients with Left Main and/or 3-Vessel Disease Undergoing Percutaneous Coronary Intervention in the Contemporary Cobalt-Chromium Everolimus-Eluting Stent Era. Korean Circ J. 2020 Jan;50(1):22-34. doi: 10.4070/kcj.2019.0097. Epub 2019 Sep 30. PMID 31642213